CLINICAL TRIAL: NCT05923034
Title: Pulmonary Infection and Clinical Pneumonia After Ischemic Stroke
Brief Title: Pulmonary Infection After Ischemic Stroke
Acronym: PICAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Other Study IDs: PICAS
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Had a Computed Tomography Scan of the Chest Within 24 Hours After Stroke Onset

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- had a computed tomography scan of the chest within 24 hours after stroke onset

SUMMARY:
To assess the frequency of signs of pulmonary infection on a chest CT and development of clinical diagnose of poststroke pneumonia，and its effect on functional outcome in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

Have a computed tomography scan of the chest within 24 hours after stroke onset

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: had a computed tomography scan of the chest within 24 hours after stroke onset
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
With radiological signs of pulmonary infection | 24 hours

SECONDARY OUTCOMES:
development of clinical poststroke pneumonia | 2 weeks or at discharge
modified Rankin Scale | 90 days

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Suzhou Municipal Hospital, Suzhou, Anhui
  - People Hospital of Rongcheng, Baoding, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - People Hospital of Ningjin, Xingtai, Hebei
  - Shihezi Municipal Hospital, Shihezi, Xinjiang
  - Xuanwu Hospital, Capital Medical University, Beijing